CLINICAL TRIAL: NCT00890162
Title: A Randomized Double-Blinded, Placebo-Controlled Study of Omalizumab for Idiopathic Anaphylaxis
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study of Omalizumab for Idiopathic Anaphylaxis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 090129; 09-I-0129
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2018-08

CONDITIONS: Anaphylaxis; Hypotension; Bronchospasm; Angioedema
Keywords: Omalizumab; Idiopathic Anaphylaxis; Serum Tryptase; Placebo-Controlled; Adult; Anaphylaxis; Allergic Reaction
MeSH Terms: conditions — Anaphylaxis; Hypotension; Bronchial Spasm; Angioedema; Hypersensitivity | interventions — Epinephrine; Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Omalizumab (Active Comparator): Subjects will receive two doses of Omalizumab while hospitalized, followed by continued outpatient therapy, every 2 to 4 weeks, for up to 6 months.
  Interventions: Drug: Epinephrine; Drug: Omalizumab (Xolair)
- Placebo (Placebo Comparator): Subjects will receive two doses of placebo while hospitalized, followed by continued outpatient therapy, every 2 to 4 weeks, for up to 6 months.
  Interventions: Drug: Epinephrine; Drug: Placebos

INTERVENTIONS:
Drug: Epinephrine
Drug: Omalizumab (Xolair)
  Arms: Omalizumab
Drug: Placebos
  Arms: Placebo

SUMMARY:
Background:

* Omalizumab is an approved drug for the treatment of asthma by the Food and Drug Administration.
* Researchers are now studying this drug in a double-blind placebo-controlled manner to assess efficacy in patients with idiopathic anaphylaxis (recurrent hypersensitive allergic episodes for which a cause is not identified).
* The study will improve understanding of the mechanisms involved in anaphylactic reactions as a response to the downregulation (a decrease in the number of receptors on the surface of cells) in mast cell (a resident cell with several types of tissues) activation, and lead to the development of strategies to better prevent or treat anaphylaxis.

Objectives:

* To determine whether treatment with omalizumab will reduce or prevent episodes of unprovoked anaphylaxis (an acute allergic reaction) in subjects with a history of idiopathic anaphylaxis.
* To assess pharmacodynamics (physiological effects of a drug) and identify patients with undiagnosed mastocytosis (rare disorders caused by too many mast cells).
* To investigate cellular and molecular mechanisms of signaling and the effect of omalizumab on mast cells or basophils (a cell in the leukocyte family that releases histamine, which affects allergic response) and explore other regulatory pathways that may be involved with modulation of mast cell degranulation.

Eligibility:

* Patients between 18 and 70 years of age who have been diagnosed with idiopathic anaphylaxis, a diagnosis that is made only after other causes of anaphylaxis have been considered.
* Patients with documented anaphylaxis episodes (mild to severe) at least six times within the past 1 year period, at least once within the last 4 months, and with at least one of the following:

  * Elevated serum tryptase above baseline within 2 hours of the event.
  * Emergency room visit with documented anaphylaxis without a known cause established by the acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (generalized hives, itching or flushing, swollen lips-tongue-throat) and at least one of the following: (1) respiratory compromise or gastrointestinal involvement (shortness of breath, wheeze-bronchospasm, throat tightness, low oxygen levels, nausea, vomiting, or abdominal pain); or (2) reduced blood pressure or associated symptoms of end-organ dysfunction (collapse, loss of consciousness, or loss of bladder or bowel control).
  * Hospitalization for anaphylaxis.
* Patients must provide a letter of referral, with copies of pertinent medical history and laboratory tests, from the prospective participant s local physician, and have the ability to give informed consent.
* Women with childbearing potential must have a negative pregnancy test, and must agree to practice abstinence or effective birth control from the start of the protocol and for 3 months following the last injection of the study drug.

Design:

* Participants will undergo a clinical evaluation, blood tests, and a bone marrow biopsy and aspirate.
* Participants will be randomized to either drug or placebo and will receive two doses of omalizumab or a matched placebo while hospitalized, followed by continued outpatient therapy, every 2 to 4 weeks, for up to 6 months.
* Participants will remain on the assigned regimen for 6 months or until they have experienced new onset of severe adverse event on one occasion within 24 hours of study medication that are related to the study drug, whichever comes first. At that time, the participant will be discontinued from drug administration.

DETAILED DESCRIPTION:
Anaphylaxis is a severe systemic reaction caused by release of mediators from mast cells and basophils. Manifestations include cutaneous, respiratory, cardiovascular, or gastrointestinal signs and symptoms. Although anaphylaxis is frequently attributed to exposure to specific foods, drugs, and insect venoms in sensitive individuals, a causative factor is not identified in 30% to 50% of patients with recurrent anaphylactic episodes (idiopathic anaphylaxis).

Currently, therapeutic options for the treatment of idiopathic anaphylaxis are limited with variable efficacy. This pilot study will examine the hypothesis that omalizumab (Xolair ) will decrease episodes of unexplained anaphylaxis in patients with idiopathic anaphylaxis. Omalizumab is approved for use in asthma. We will examine the safety profile and efficacy of omalizumab in patients with anaphylaxis. In addition, the study will investigate whether patients with anaphylaxis have unique molecular and cellular defects in mast cells that result in these cells being more susceptible to degranulation.

The study will enroll patients with idiopathic anaphylaxis. Patients will undergo a clinical evaluation, blood tests, and a bone marrow biopsy and aspirate. Patients will be randomized to either drug or placebo and will receive, in a double-blind placebo-controlled approach, 2 doses of omalizumab or a matched placebo while hospitalized, followed by continued outpatient therapy, every 2 to 4 weeks, for up to 6 months. Patients will remain on the assigned regimen if they have experienced anaphylactic events (post 24-hr window) determined to be unrelated to study drug or have been followed for 6 months, whichever comes first. These unrelated events would be determined by the PI not to jeopardize patient safety or restrict the use of additional therapy such as corticosteroids to control symptoms. After this point, the patient may be discontinued from drug administration until unblinding. This design ensures that no patient will have anaphylactic episodes while on placebo if other therapy is medically indicated. Research studies will be conducted to elucidate other markers or pathways of mast cell regulation.

The primary outcome will be a reduction in the number and timing of anaphylactic events during the randomized phase. Secondary outcomes will include a reduction in surface IgE receptors on basophils, identification of mutations in c-kit, and evaluation of the efficacy of omalizumab on other mediator-induced symptoms associated with anaphylaxis. The study will improve the understanding of the mechanisms involved in anaphylactic reactions as a response to the downregulation of mechanisms involved in mast cell activation that could, in turn, lead to development of strategies to better prevent or treat anaphylaxis.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers must satisfy all of the following inclusion criteria to be eligible for this study.

Subject must be at least 18 years of age and no older than 70 years of age.

Diagnosis of idiopathic anaphylaxis, a diagnosis of exclusion, assigned after other causes of anaphylaxis and other diseases in the differential diagnoses have been considered.

Anaphylaxis episodes (mild-severe) at least 6 times within the past 1 year period, documented according to medical records physician report, or patient report and 1 episode within the last 4 months, and with at least 1 of the following:

1. Elevated serum tryptase above baseline within 2 hours of the event.
2. Emergency room visit with documented anaphylaxis without an etiology established by the acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (e.g., generalized hives, pruritus or flushing, swollen lips-tongue-uvula) [Grade 1]* and at least 1 of the following:

   1. Respiratory compromise or gastrointestinal involvement (e.g., dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow, hypoxemia, nausea, vomiting, or abdominal pain [Grade 2]*).
   2. Reduced blood pressure or associated symptoms of end-organ dysfunction (e.g., hypotonia [collapse], syncope, or incontinence [Grade 3]*).
3. Hospitalization for anaphylaxis: hospital records with documented anaphylaxis without known cause established by the acute onset of an illness (minutes to several hours) with involvement of the skin, mucosal tissue, or both (e.g., generalized hives, pruritus or flushing, swollen lips-tongue-uvula) [Grade 1]*) and at least one of the following:

   1. Respiratory compromise or gastrointestinal involvement (e.g., dyspnea, wheeze-bronchospasm, stridor, reduced peak expiratory flow, hypoxemia, nausea, vomiting, or abdominal pain [Grade 2]*).
   2. Reduced blood pressure or associated symptoms of end-organ dysfunction (e.g., hypotonia [collapse], syncope, or incontinence [Grade 3]*).
4. Letter of referral, with copies of pertinent medical history and laboratory tests, from prospective study participant s local physician.
5. Ability to give informed consent.
6. Women of childbearing potential must have a negative beta-HCG serum or urine pregnancy test prior to each injection, and must agree to practice abstinence or effective contraception from initiation of the protocol and for 3 months following the last infusion of the study agent (effective contraception methods include abstinence; surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap, or sponge; or hormonal contraception).

   * Severity grading of anaphylaxis

EXCLUSION CRITERIA:

A volunteer who satisfies any of the following exclusion criteria will be ineligible to participate in this study.

1. Presence of conditions which, in the judgment of the investigator or the referring physician, may put the subject at undue risk for study participation or travel (such as an acute infection, severe thrombocytopenia, coronary artery disease, uncontrolled hypertension, congestive heart failure, chronic beta blocker therapy such as atenolol or metoprolol, or myeloproliferative disease).
2. History of malignancy
3. Known cause for anaphylaxis or flushing
4. Diagnosis of mastocytosis
5. Inability to provide informed consent
6. Inability or refusal to undergo a bone marrow biopsy and aspirate
7. HIV positive or other known immunodeficiency
8. Active or chronic hepatitis
9. Use of any other investigational agent within 30 days of the study
10. Current use of chronic-oral corticosteroids or other immunosuppressant medications
11. Pregnant or nursing women
12. Positive pregnancy test
13. IgE levels and subject s weight that cause dosing to be above dosing guidelines.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04-27; Primary Completion 2018-07-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melody C Carter, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Thong BY, Cheng YK, Leong KP, Tang CY, Chng HH. Anaphylaxis in adults referred to a clinical immunology/allergy centre in Singapore. Singapore Med J. 2005 Oct;46(10):529-34. PMID 16172772
- [Background] Webb LM, Lieberman P. Anaphylaxis: a review of 601 cases. Ann Allergy Asthma Immunol. 2006 Jul;97(1):39-43. doi: 10.1016/S1081-1206(10)61367-1. PMID 16892779
- [Background] Neugut AI, Ghatak AT, Miller RL. Anaphylaxis in the United States: an investigation into its epidemiology. Arch Intern Med. 2001 Jan 8;161(1):15-21. doi: 10.1001/archinte.161.1.15. PMID 11146694
- [Background] Carter MC, Robyn JA, Bressler PB, Walker JC, Shapiro GG, Metcalfe DD. Omalizumab for the treatment of unprovoked anaphylaxis in patients with systemic mastocytosis. J Allergy Clin Immunol. 2007 Jun;119(6):1550-1. doi: 10.1016/j.jaci.2007.03.032. Epub 2007 May 3. No abstract available. PMID 17481708
- [Background] Constantine GM, Bressler PB, Petroni D, Metcalfe DD, Carter MC. Twelve-year follow-up of omalizumab therapy for anaphylaxis in 2 patients with systemic mastocytosis. J Allergy Clin Immunol Pract. 2019 Apr;7(4):1314-1316. doi: 10.1016/j.jaip.2018.07.041. Epub 2018 Aug 24. No abstract available. PMID 30149096
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-I-0129.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omalizumab | Placebo
Started | 8 | 8
Completed | 6 | 7
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Reduction in the Number and Timing of Anaphylactic Events in Subjects With a History of Frequent Idiopathic Anaphylaxis.
Description: To determine if treatment with omalizumab over 6 months will produce a reduction in the number and timing of anaphylactic events in subjects with a history of frequent idiopathic anaphylaxis. Ordinal outcome of participants based on number of events in 6 months after baseline and timing of first event. Events were calculated based on detailed event logs maintained by the patients and collected every 2-4 weeks based on injection schedule. Mean percent change in number of events experienced while on study agent for each subject and results presented as a group.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of change of events
Arm/Group | Omalizumab | Placebo
Number analyzed (Participants) | 8 | 8
percentage of change of events | 32 [6 to 57] | 6 [-38 to 50]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Omalizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=8) | Placebo (N=8)
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (N=8) | Placebo (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Chest discomfort (Cardiac disorders) | 1 | 0
Chest pain (Cardiac disorders) | 1 | 0
Dizziness (Cardiac disorders) | 1 | 2
Dyspnoea (Cardiac disorders) | 2 | 1
Pulmonary congestion (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Syncope (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Hypoglycaemia (Endocrine disorders) | 2 | 0
Polydipsia (Endocrine disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Seasonal allergy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Oral candidiasis (Gastrointestinal disorders) | 0 | 1
Oropharyngeal pain (Gastrointestinal disorders) | 2 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Flushing (General disorders) | 2 | 1
Injection site pain (General disorders) | 6 | 6
Injection site pruritus (General disorders) | 1 | 0
Injection site reaction (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Hypoalbuminaemia (Hepatobiliary disorders) | 1 | 0
Urticaria (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dysphonia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Personality change (Nervous system disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Although we received multiple inquiries for this study, it was difficult to find subjects who met all eligibility criteria and who were also willing to participate in a double-blind placebo-controlled trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT00890162/Prot_SAP_000.pdf